CLINICAL TRIAL: NCT06552351
Title: Needle-Free Jet Injection Versus Traditional Lidocaine Needle Infiltration for Local Anesthesia in Infant Lumbar Puncture
Brief Title: Needle-Free Lidocaine Injection vs Traditional Local Anesthesia in Infant Lumbar Puncture
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17204
Record Dates: First submitted 2024-07-29; First posted 2024-08-14 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Anesthesia
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to receive either needle-free jet injection or traditional lidocaine needle infiltration for local anesthesia during infant lumbar puncture
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Needle-Free Jet Injection of 1 % lidocaine (Experimental): Device: Needle-Free Jet Injection The needle-free jet injection device delivers 1 % Lidocaine through high-pressure fluid without the use of a needle. This method aims to reduce the pain associated with needle-based anesthesia during infant lumbar punctures.
  Other Names:
  • Jet Injection Device, J-tip
  Interventions: Device: Needle-Free Jet Injection of 1 % lidocaine
- Traditional needle infiltration of 1% lidocaine (Experimental): Traditional needle infiltration involves injecting 1% lidocaine with a needle to provide local anesthesia before an infant lumbar puncture. This method is the standard practice for pain management in such procedures.
  Other Names:
  • traditional needle infiltration of 1% lidocaine
  Interventions: Other: traditional needle infiltration of 1% lidocaine

INTERVENTIONS:
Device: Needle-Free Jet Injection of 1 % lidocaine — The needle-free jet injection device delivers 1% lidocaine through high-pressure fluid without the use of a needle. This method aims to reduce the pain associated with needle-based anesthesia during infant lumbar punctures.
  Other Names: Jet Injection Device, J-tip injection of 1 % lidocaine
  Arms: Needle-Free Jet Injection of 1 % lidocaine
Other: traditional needle infiltration of 1% lidocaine — Traditional needle infiltration involves injecting 1% lidocaine with a needle to provide local anesthesia before an infant lumbar puncture. This method is the standard practice for pain management in such procedures.
  Arms: Traditional needle infiltration of 1% lidocaine

SUMMARY:
We hypothesize that the J-Tip needle-free jet-injection system offers comparable pain control and greater provider satisfaction due to its less invasive nature compared to traditional needle infiltration of 1% lidocaine in infants undergoing lumbar punctures.

Our aim is to evaluate the efficacy and feasibility of different local anesthetic techniques in the ED setting by comparing traditional lidocaine needle infiltration with J-tip.

DETAILED DESCRIPTION:
Lumbar punctures (LPs) play a key role in diagnosing meningitis in febrile infants. The use of local anesthesia is critical to the success of these procedures. Traditional anesthesia techniques, including needle injections and the application of topical anesthetic creams, have been effective in managing pain and enhancing the outcomes of LPs. Recently, the introduction of needle-free jet injection technology, such as the J-Tip system, offers a quicker and less invasive method for delivering local anesthesia.

This research compares the effectiveness of the J-Tip with that of traditional 1% lidocaine infiltration for local anesthesia during LPs in infants.

The investigators hypothesize that the J-Tip needle-free jet-injection system offers comparable pain control and greater provider satisfaction due to its less invasive nature compared to traditional needle infiltration of 1% lidocaine in infants undergoing lumbar punctures.

The aim is to evaluate the efficacy and feasibility of different local anesthetic techniques in the ED setting by comparing traditional 1% lidocaine needle infiltration with administration of 1% lidocaine the J-Tip.

Secondary outcomes include the number of attempts to successfully perform the LP, perceptions of pain management effectiveness by ED providers, the need for additional lidocaine, skin condition at the LP site, and the overall success rate of the LP procedures.

EXPERIMENTAL DESIGN:

A single-center, randomized, controlled trial will compare the efficacy of J-Tip-injected lidocaine with conventional needle-injected lidocaine in providing anesthesia for infants undergoing lumbar punctures.

PROPOSED PROCEDURE:

Infants aged 0 to 3 months presenting to the Oklahoma Children's Hospital Emergency Department between July 1, 2024, through June 30, 2025, who require an LP as part of their ED evaluation will be recruited.

Randomization Strategy:

Participants who consent will be randomly divided into two groups: one receiving local anesthesia via the J-Tip syringe containing 1% lidocaine (experimental group) and the other through needle infiltration with the same concentration of lidocaine (control group). Randomization assignments will be provided in sealed envelopes and kept with the study team to be included in a study packet along with the consent forms to be reviewed at the time of enrollment.

The ED provider performing the LP will independently evaluate pain levels using the Neonatal Infant Pain Scale (NIPS) immediately before the LP begins and at the time of needle insertion.

A brief period of up to 5 minutes will follow the topical anesthesia application to allow infants to calm and reach a steady state, accounting for any initial discomfort or startle response.

After the LP, attending providers will complete a questionnaire detailing the number of attempts, any encountered difficulties, additional lidocaine usage, their assessment of pain control during the procedure, any skin changes at the LP site, and LP success, defined as obtaining cerebrospinal fluid.

Outcome Measures:

Primary Outcome: Pain levels, as measured by NIPS scores, immediately before the LP and at needle insertion.

The NIPS (Neonatal Infant Pain Scale) is a scoring system used to assess pain in newborns and infants up to 1 year of age. It is a behavioral scale that evaluates specific criteria to determine the level of pain the infant may be experiencing.

NIPS Scoring System:

Facial Expression (0-1 points) 0: Relaxed facial expression

1: Grimace Cry (0-2 points) 0: No cry

1. Whimper
2. Vigorous cry Breathing Patterns (0-1 points)

0: Relaxed breathing

1: Change in breathing patterns (e.g., irregular, fast, or slow breathing) Arm Movements (0-1 points) 0: Relaxed, no movement or only gentle movements

1: Flexed or extended movements (restless, jerking) Leg Movements (0-1 points) 0: Relaxed, no movement or only gentle movements

1: Flexed or extended movements (restless, jerking) State of Arousal (0-1 points) 0: Sleeping or calm

1: Fussy

Scoring Interpretation:

0-2 points: Mild or no pain 3-4 points: Moderate pain 5-7 points: Severe pain

Secondary Outcomes: Include the number of LP attempts, any difficulties encountered (open-ended), provider's perception of pain control (1-5 scale), additional lidocaine use, post-procedure skin reactions (classified as minor/moderate or severe induration, bleeding), and LP success. Additionally, it will be determined if the LP was traumatic by reviewing patient charts, defined as having a cerebrospinal fluid (CSF) red blood cell (RBC) count of ≥ 1000 cells/mm³.

Provider Information: Details about the providers performing the LP, including their level of training (APP, fellow, attending, resident) and prior experience with LPs (categorized as 0-5, 6-10, 11-20, >20 attempts), will be documented.

Data will be entered into REDCap and only authorized key study personnel will have access. Identifiers will be removed, and the de-identified information may be used for future research without additional informed consent from the participant.

ELIGIBILITY:
Infants requiring lumbar puncture for diagnostic or therapeutic purposes

* Age 0 to 3 months
* Parental/guardian consent obtained

Exclusion Criteria:

* Infants with known allergy or hypersensitivity to lidocaine or components of the needle-free jet injection device
* Infants with significant skin infection or dermatitis at the site of injection
* Infants with coagulopathy or any bleeding disorder
* Infants with any other condition that, in the opinion of the investigator, would make participation in the study unsafe or not in the best interest of the infant

Ages: 1 Day to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Pain Score | Immediately post-procedure (within 5 minutes after the lumbar puncture)
  The primary outcome measure will be the pain score of infants undergoing lumbar punctures, assessed using a validated pain scale appropriate for infants.
Procedure Success Rate | During the procedure
  The success rate of the lumbar puncture procedure, defined as obtaining an adequate CSF sample on the first attempt without the need for additional anesthesia.
Caregiver Satisfaction | Within 1 hour post-procedure
  Caregiver satisfaction with the anesthesia method used, measured using a standardized survey or questionnaire completed after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Laughy, MD, Principal Investigator — University of Oklahoma
Locations (1):
- Oklahoma Children's Hospital, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Baxter AL, Welch JC, Burke BL, Isaacman DJ. Pain, position, and stylet styles: infant lumbar puncture practices of pediatric emergency attending physicians. Pediatr Emerg Care. 2004 Dec;20(12):816-20. doi: 10.1097/01.pec.0000148030.99339.fe. PMID 15572969
- [Background] Caltagirone R, Raghavan VR, Adelgais K, Roosevelt GE. A Randomized Double Blind Trial of Needle-free Injected Lidocaine Versus Topical Anesthesia for Infant Lumbar Puncture. Acad Emerg Med. 2018 Mar;25(3):310-316. doi: 10.1111/acem.13351. Epub 2017 Dec 26. PMID 29160002
- [Background] Use of Jet-Injected Lidocaine to Reduce Venipuncture Pain. AAP Grand Rounds, 2016. 35(2): p. 13-13.
- [Background] Hajimaghsoudi M, Vahidi E, Momeni M, Arabinejhad A, Saeedi M. Comparison of local anesthetic effect of lidocaine by jet injection vs needle infiltration in lumbar puncture. Am J Emerg Med. 2016 Jul;34(7):1225-9. doi: 10.1016/j.ajem.2016.03.030. Epub 2016 Mar 16. PMID 27055606
- [Background] Nigrovic LE, Kuppermann N, Neuman MI. Risk factors for traumatic or unsuccessful lumbar punctures in children. Ann Emerg Med. 2007 Jun;49(6):762-71. doi: 10.1016/j.annemergmed.2006.10.018. Epub 2007 Feb 23. PMID 17321005
- [Background] Fein D, Avner JR, Khine H. Pattern of pain management during lumbar puncture in children. Pediatr Emerg Care. 2010 May;26(5):357-60. doi: 10.1097/PEC.0b013e3181db2026. PMID 20404782
- [Background] Ferayorni A, Yniguez R, Bryson M, Bulloch B. Needle-free jet injection of lidocaine for local anesthesia during lumbar puncture: a randomized controlled trial. Pediatr Emerg Care. 2012 Jul;28(7):687-90. doi: 10.1097/PEC.0b013e31825d210b. PMID 22743744
- [Background] Hoyle JD Jr, Rogers AJ, Reischman DE, Powell EC, Borgialli DA, Mahajan PV, Trytko JA, Stanley RM. Pain intervention for infant lumbar puncture in the emergency department: physician practice and beliefs. Acad Emerg Med. 2011 Feb;18(2):140-4. doi: 10.1111/j.1553-2712.2010.00970.x. PMID 21314772